CLINICAL TRIAL: NCT06189456
Title: Evaluation of the Efficacy and Safety of Eye Drops With Hyaluronic Acid Sodium Salt 0.30% and Amino Acid (BLUgel A Free) in Patients With Moderate to Severe Dry Eye Syndrome and Hyaluronic Acid Sodium Salt 0.15% and Amino Acid (BLUyal A Free) in Patients With Mild Dry Eye Syndrome
Brief Title: Evaluation of Performance and Safety of Eye Drops With Hyaluronic Acid 0.30% and 0.15%
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS01-21-01
Record Dates: First submitted 2023-12-01; First posted 2024-01-03 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Syndrome (DES)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: profit, multicentric, prospective, open-label, non-pharmacological clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients with diagnosis of moderate to severe dry eye syndrome will start a 60 days treatment period with BLUgel A free (2 drops per eye, 3 times a day, bilaterally)
  Interventions: Device: BLUgel A
- Group B (Experimental): Patients with diagnosis of mild dry eye syndrome will start a 60 days treatment period with BLUyal A free (2 drops per eye, 3 times a day, bilaterally).
  Interventions: Device: BLUyal A

INTERVENTIONS:
Device: BLUgel A — BLUgel A: Hyaluronic Acid Eye Drops 0.30%
  Arms: Group A
Device: BLUyal A — BLUyal A:Hyaluronic Acid Eye Drops 0.15%
  Arms: Group B

SUMMARY:
This is a profit, multicentric, prospective, open-label, non-pharmacological clinical investigation aim to evaluate the efficacy and tollerability of two types of eye drops containing Hyaluronic acid (HA) with different concentration as 0.30% (BLUgel A) and 0.15% (BLUyal A). the study will consider patients affected by moderate to severe dry eye syndrome which will be treated with HA 0.30% while patients affected by mild dry eye syndrome will be treated with HA 0.15%.Dry eye syndrome (DES) is defined as a multifactorial disease of the ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface.Based on the available background on the use of HA in the management of DES, this investigation has been designed to assess the efficacy of HA- and amino acid-based product BLUgel A free and BLUyal A free, in patients with moderate to severe and mild dry eye syndrome, respectively.

DETAILED DESCRIPTION:
This is a profit, multicentric, prospective, open-label, non-pharmacological clinical investigation. Patients will have an initial screening/baseline Visit 1-T0 (day 0). Patients with diagnosis of moderate to severe dry eye syndrome will start a 60 days treatment period with BLUgel A free (2 drops per eye, 3 times a day, bilaterally), while patients with diagnosis of mild dry eye syndrome will start a 60 days treatment period with BLUyal A free (2 drops per eye, 3 times a day, bilaterally).

The following on-site visits will be performed: Visit 2-T1 (day 15 [+3]), Visit 3-T2 (day 30 [+3]) and Visit 4-T3 (day 60 [+3]). Visit 3-T2 and Visit 4-T3 should be performed preferably at day 30 and day 60 respectively. In case Visit 3-T2 is postponed within the allowed window, treatment has to be continued by the patient without interruption.

A total of 100 male or female patients who have been diagnosed with mild or moderate to severe dry eye syndrome are planned to be enrolled. Dry eye syndrome will be classified according to Tear Film and Ocular Surface Society (TFOS) Dry Eye Workshop (DEWS) (2007 version) definition. Patients with diagnosis of moderate to severe dry eye syndrome will be treated with BLUgel A free for 60 days, patients with diagnosis of mild dry eye syndrome will be treated BLUyal A free for 60 days. Patients will be stratified in the two categories of severity, i.e. 50 patients with moderate/severe dry eye syndrome treated with BLUgel A free and 50 patients with mild dry eye syndrome treated with BLUyal A free.

Patients are not permitted to use a concomitant drug or device interfering with the dryness of the eye, such as corticosteroid and antibiotic eye drops; instead, they are permitted to use any drug or device non-interfering with the treatment of dry eye syndrome and not affecting the effectiveness of BLUgel A free or BLUyal A free or the occurrence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria at the screening/baseline visit will be considered as eligible for the investigation:

1. Patients having signed written informed consent to participate in the investigation obtained according to Good Clinical Practice (GCP);
2. Patients having an age ≥ 18 years;
3. Patients with diagnosis of dry eye syndrome (according to Tear Film and Ocular Surface Society [TFOS] Dry Eye Workshop [DEWS] definition);
4. Diagnosis of dry eye syndrome for the investigation assessed through at least the following exams: slit lamp examination (SLE), tear (lacrimal) meniscus exam, Schirmer's test I, TFBUT, cornea and conjunctiva staining, IDEEL questionnaire ("Dry Eye Symptom-Bother" module); 4a) Diagnosis of mild dry eye syndrome will be based on the following criteria:

   * TFBUT 7-10 sec
   * Schirmer's test I 7-10 mm
   * Fluorescein staining of the cornea and conjunctiva (NEI scale value) <7
   * IDEEL questionnaire ("Dry Eye Symptom-Bother" module) score 40-50
   * Patient not treated in the previous 15 days for dry eye syndrome 4b) Diagnosis of moderate to severe dry eye syndrome will be based on the following criteria:
   * TFBUT < 7 sec
   * Schirmer's test I < 7 mm
   * Fluorescein staining of the cornea and conjunctiva (NEI scale value) ≥7
   * IDEEL questionnaire ("Dry Eye Symptom-Bother" module) score >50
   * Dry eye syndrome treatment permitted; no ophthalmic gel treatment permitted

   In case of bilateral dry eye syndrome, both eyes will be treated but only the worst eye, defined as the eye with the higher severity of impairment according to the Investigator's judgment based on the above exams, will be considered for assessments (although both eyes will be treated). In the case of bilateral dry eye syndrome with both eyes having the same level of impairment, the right eye will be considered for assessments by convention; In case of monolateral dry eye syndrome, both eyes will be treated. Evaluations of both the eyes will be collected but only target eye evaluations will be used for statistical analysis.
5. Patients being able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and patients able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on Investigator's judgment;
6. Female patients having a negative urine pregnancy test result at screening and using an appropriate method of contraception for at least 30 days before inclusion and during the whole investigation period, according to the definition of Note 3 of ICH M3 Guideline*, if females of childbearing potential (i.e., not permanently sterilized - post hysterectomy or tubal ligation status - or not postmenopausal);

   * Note: According to the definition of Note 3 of ICH M3 Guideline a highly effective method is defined as those which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Highly effective birth control methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

Patients who fulfil any of the following criteria at the screening/baseline visit will be excluded from the investigation:

1. Patients with mild dry eye syndrome that have used eye drops product in the 15 days preceding the screening/baseline visit.

   Patients with moderate to severe dry eye syndrome may have used treatment for dry eye syndrome in the 15 days preceding the screening/baseline visit, with the exception of gel compounds;
2. Patients under treatment with corticosteroids or antibiotics eye drops, hypotony-inducing products or any other therapy that, as per Investigator's opinion, could interfere with the assessment of the efficacy or incidence of adverse events;
3. Patients with presence or history of any systemic or ocular disorder, condition or disease (with particular attention to malignancies and neuro-oncological diseases) that, according to Investigator's judgment, can interfere with the conduct of the required investigation procedures or the assessment of the efficacy or the interpretation of the investigation results or the incidence of adverse events;
4. Patients with glaucoma;
5. Patients that use therapeutic or refractive contact lenses;
6. Patients with hypersensitivity and/or allergy to any of the BLUgel A free or BLUyal A free ingredients;
7. History of ocular surgery in either eye, excluding corneal refractive or cataract procedures, within 90 days of investigation enrolment;
8. Patients not being able to apply during the investigation any eye drops product;
9. Patients treated with antidepressant, antiepileptic, antihistamine, anticholinergic drug;
10. Patients participating to another clinical study/investigation at the same time as the present investigation or within 30 days;
11. Patients who have history of drug, medication or alcohol abuse or addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessment from baseline | Day 30
  -Changes from baseline (T0) to Day 30 (T2) of overall score of National Eye Institute (NEI) corneal (range 0-15) and conjunctival (range 0-18) fluorescein staining, following treatment with BLUgel A free ophthalmic solution in patients with moderate to severe dry eye syndrome;
Changes in Tear Film Break-Up Time (TFBUT) from baseline | Day 30
  - Changes from baseline (T0) to Day 30 (T2) in Tear Film Break-Up Time (TFBUT) values, following treatment with BLUyal A free ophthalmic solution in patients with mild dry eye syndrome. The TFBUT will be measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differ by more than 2 seconds a third reading will be taken. The TFBUT value will be the average of the 2 or 3 measurements.

SECONDARY OUTCOMES:
Efficacy Assessment from baseline in patients with moderate to severe dry eye syndrome | Day 60
  Change from baseline (T0) to Day 60 (T3) of overall score of NEI corneal (range 0-15) and conjunctival fluorescein (range 0-18) staining following treatment with BLUgel A free, and change from baseline (T0) to Day 30 (T2) and Day 60 (T3) of overall score of NEI corneal and conjunctival fluorescein staining following treatment with BLUyal A free ophthalmic solution. the maximum score of the sum of NEI corneal and conjunctival total score is 33.
Efficacy Assessment from baseline | Day 30 and Day 60
  * Changes from baseline (T0) to Day 30 (T2) and Day 60 (T3) in Tear Film Break-Up Time (TFBUT) values, following treatment with BLUgel A free ophthalmic solution in patients with mild dry eye syndrome.
  * Changes from baseline (T0) to Day 60 (T3) in Tear Film Break-Up Time (TFBUT) values, following treatment with BLUyal A free ophthalmic solution in patients with mild dry eye syndrome.
  The TFBUT will be measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differ by more than 2 seconds a third reading will be taken. The TFBUT value will be the average of the 2 or 3 measurements.
Efficacy Assessment from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in non-invasive Break-Up Time (niBUT) measured via Tearcheck®, following treatment with BLUgel A free, and with BLUyal A free ophthalmic solution. niBUT evaluates the stability and the break-up time of the tear film. In particular, niBUT shows site and time of ruptures of the tear film. During a 10-second imaging, Tearcheck® evaluates the tear film surface 3 times per second. For better readability, results are then grouped into 2-second increments. niBUT will be expressed in seconds.
Change in non-invasive Break-Up Time (niBUT) from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in non-invasive Break-Up Time (niBUT) measured via Tearcheck®, following treatment with BLUgel A free, and with BLUyal A free ophthalmic solution. niBUT evaluates the stability and the break-up time of the tear film. In particular, niBUT shows site and time of ruptures of the tear film. During a 10-second imaging, Tearcheck® evaluates the tear film surface 3 times per second. For better readability, results are then grouped into 2-second increments. niBUT will be expressed in seconds.
Assessment of Tear meniscus height after treatment compared to baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) of conjunctival, measured via Tearcheck®, following treatment with BLUgel A free and with BLUyal A free ophthalmic solution.
  The Tearcheck® instrument will be used to measure niBUT, tear meniscus height, conjunctival hyperaemia and meibography, which will not be performed at Visit 2-T1 (Day 15 +3); all the remaining parameters will be measured at any visit.
  The tear meniscus will be evaluated in the lower eyelid and shows, if there is sufficient tear production before the next eye blink. Two values will be calculated: 1) tear meniscus measurement below iric centre; 2) thickest measurement of the tear meniscus. The tear meniscus height will be expressed in millimetres.
Assessment of conjunctival hypaermia from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in conjunctival hypaermia, measured via Tearcheck®, following treatment with BLUgel A free and with BLUyal A free ophthalmic solution. niBUT evaluates the stability and the break-up time of the tear film.The Tearcheck® instrument will be used to measure niBUT, tear meniscus height, conjunctival hyperaemia and meibography, which will not be performed at Visit 2-T1 (Day 15 +3); all the remaining parameters will be measured at any visit.
Assessment of possible changes in meibomian gland from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in meibography, measured via Tearcheck®, following treatment with BLUgel A free and with BLUyal A free ophthalmic solution. Meibography makes it possible to visualize the meibomian glands. This visualization is useful in explaining the anatomical structure responsible for the production of the lipid film to the patient. The result will be expressed as percentage of loss of glands compared to an individual with all of the glands present.
Assessment of total tear secretion from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in Schirmer's Test I values following treatment with BLUgel A free and with BLUyal A free ophthalmic solution.
  The Schirmer's test I (Schirmer, 1903) measures the quantity of total tear secretion, including reflex and basal tears, which are produced by the eye. A 35 mm x 5 mm size filter paper strip is used to measure the amount of tears that are produced over a period of 5 minutes. Without instilling anaesthetic drops, the Schirmer strips are inserted into the eye under the eyelid and into the lower conjunctival fornix near the lateral corner, avoiding contact with the cornea. The paper strip remains in the conjunctival fornix for 5 minutes to measure the production of tears. The wet portion of the strip is measured in millimetres. The test is done under ambient light. The patient is instructed to look forward and to blink normally during the course of the test.
Assessment of impact of Dry Eye on Everyday Life (IDEEL) from baseline | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T2) and Day 60 (T3) in score of Impact of Dry Eye on Everyday Living (IDEEL) questionnaire ("Dry Eye Symptom-Bother" module) following treatment with BLUgel A free and with BLUyal A freeophthalmic solution. The Impact of Dry Eye on Everyday Life (IDEEL) questionnaire is a comprehensive dry eye specific questionnaire developed to evaluate symptom-related bother, impact on daily life and treatment satisfaction in a population with dry eye (Abetz et al, 2011). There are 57 items grouped into 3 different modules: i) the Dry Eye Impact on Daily Life" (3 section: daily living activities (9 items), emotional impact (12 items) and impact of work (6 items); ii) the "Dry Eye Symptom-Bother" (20 items), and iii) the "Dry Eye Treatment Satisfaction" (10 items). Only the "Dry Eye Symptom-Bother" (10 items) will be evaluated in this investigation
Incidence and nature of treatment-emergent adverse events | Day 30 and Day 60
  Incidence and nature of treatment-emergent adverse events (TEAEs) as well as of the treatment-emergent serious adverse events (TESAEs); Incidence and nature of the Adverse Device Effects (ADEs); Incidence and nature of the Serious Adverse Device Effects (SADEs); Incidence and nature of Investigational Medical Device Deficiencies (IMDDs)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mencucci, MD, Principal Investigator — AOU Careggi
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria-Renato Dulbecco, Catanzaro, CZ
  - AOU Careggi, Florence
  - ASST Santi Paolo e Carlo P.O San Paolo, Milan

IPD SHARING:
Plan to Share IPD: No